CLINICAL TRIAL: NCT07132632
Title: Effect of a Multicomponent Therapeutic Exercise Program in Primary Care on Frailty and Sarcopenia in Older Adults
Acronym: FRACTEP-65
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Yaiza Casas, Principal Investigator and Physiotherapist, Primary Care - Institut Català de la Salut (ICS), Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IDIAP-FRAIL65
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Sarcopenia; Aging; Exercises Therapy
MeSH Terms: conditions — Frailty; Sarcopenia | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Multicomponent Exercise Intervention
  Interventions: Behavioral: 12-week multicomponent therapeutic exercise program including supervised and home-based sessions focused on strength, balance, mobility, and aerobic capacity
- Control Arm (Placebo Comparator)
  Interventions: Behavioral: Placebo Pre-Treat

INTERVENTIONS:
Behavioral: 12-week multicomponent therapeutic exercise program including supervised and home-based sessions focused on strength, balance, mobility, and aerobic capacity — This intervention consists of a 12-week multicomponent therapeutic exercise program for older adults with mild to moderate frailty. Participants will complete 12 sessions (8 supervised in primary care and 4 home-based), each lasting approximately 60 minutes. Sessions include warm-up, strength exercises (using body weight or elastic bands), moderate aerobic activity (e.g., walking or pedaling), balance and coordination training (including dual tasks), and a cool-down phase. The program follows FITT-VP principles and is tailored to functional capacity. Intensity is monitored using the Borg scale (CR10 and RPE), estimated 1RM (20-80%), and 64-76% HRmax. Exercises are progressively adjusted in volume, intensity, and complexity. Home sessions are guided by an illustrated manual and reinforced by biweekly follow-up phone calls to promote adherence and safety. The intervention is aligned with international guidelines and aims to improve physical performance, reduce frailty and sarcopenia.
  Arms: Arm 1
Behavioral: Placebo Pre-Treat — The pre-intervention period (Month 0 to Month 3) will serve as the control phase, during which participants will receive no specific exercise program. From Month 3 to Month 6, the intervention phase will begin. Participants act as their own control.
  Arms: Control Arm

SUMMARY:
Background:

Frailty and sarcopenia are common conditions in older adults that increase the risk of disability, dependence, and hospitalizations. Frailty is characterized by decreased physiological reserve and functional capacity, while sarcopenia refers to the loss of muscle mass, strength, and performance. Both conditions are prevalent among older adults and represent a growing public health challenge as the population ages.

Objective:

This study aims to evaluate the effectiveness of a multicomponent therapeutic exercise program in reducing frailty and improving clinical parameters related to sarcopenia in community-dwelling older adults aged 65 years or older who attend primary care centers.

Study Design:

This is a quasi-experimental, multicenter, single-group pre-post clinical trial. The study includes two phases: a control phase (pre-intervention observation) and an experimental phase (intervention). Each participant will act as their own control.

Participants:

60 older adults aged 65 or older will be recruited from primary care centers in the Baix Llobregat region (Catalonia, Spain). Eligibility criteria include mild to moderate frailty (Clinical Frailty Scale 4-6), ability to walk independently (with or without a walking aid), cognitive ability to follow instructions (MMSE ≥ 20), and clinical stability. Exclusion criteria include severe frailty, major cognitive impairment, acute illness, or participation in another structured exercise program.

Intervention:

Participants will take part in a 12-week multicomponent exercise program including 8 supervised sessions at the primary care center and 4 home-based sessions. Each session will last 60 minutes and include strength training, balance exercises, aerobic activity, and flexibility. The program follows FITT-VP principles (frequency, intensity, time, type, volume, and progression). Home sessions will be supported with illustrated manuals and biweekly follow-up calls.

Outcomes:

The primary outcome is the change in frailty level measured by the Clinical Frailty Scale (CFS). Secondary outcomes include handgrip strength, SARC-F score, Short Physical Performance Battery (SPPB), 4-meter walk test, Timed Up and Go (TUG), muscle mass index, rectus femoris and vastus lateralis ultrasound, cognitive status (MMSE), nutritional status (MNA-SF), falls, and hospitalizations. Assessments will be conducted at baseline (month 0), after the control phase (month 3), and after the intervention (month 6).

Significance:

This study will provide evidence on the medium-term effectiveness of a short, structured, and feasible intervention implemented in real-life primary care settings. If effective, this program could be integrated into preventive strategies to reduce frailty and sarcopenia, promote autonomy, and improve the quality of life among older adults. Results will inform clinical guidelines and contribute to the development of scalable interventions for aging populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older, receiving care from primary care physiotherapists at participating health centers.
* Clinical Frailty Scale (CFS) score between 4 and 6 (indicating vulnerable, mild, or moderate frailty).
* Ability to walk independently, with or without assistive devices (excluding habitual wheelchair use).
* Clinically stable, defined as the absence of acute events or clinical decompensation in the previous 4 weeks.
* Sufficient cognitive ability to understand and follow basic instructions, or the availability of an actively involved caregiver (MMSE ≥ 20 or equivalent).
* Signed informed consent from the participant or their legal representative.

Exclusion Criteria:

* Diagnosis of severe frailty or advanced dependence (CFS ≥ 7).
* Severe neurological or musculoskeletal disorders that limit safe exercise participation (e.g., Parkinson's disease, stroke with major sequelae, disabling arthropathies).
* Uncontrolled cardiac, respiratory, or other medical conditions that contraindicate physical activity.
* Moderate to severe cognitive impairment, defined by MMSE < 20 or a clinical diagnosis of dementia with significant functional limitations.
* Simultaneous participation in other structured physical intervention programs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-02 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Frailty Scale (CFS) Score at 6 Months | Baseline (Month 0) to Month 6
  Clinical Frailty Scale (CFS) is a 9-point ordinal scale assessing functional and clinical status in older adults. A change of ≥0.5 points is considered clinically significant.

SECONDARY OUTCOMES:
Baseline (Month 0) to Month 6 | Baseline (Month 0) to Month 6
  Handgrip strength measured using a Jamar® dynamometer. The average of three trials per hand will be used. A decrease indicates lower muscle strength, a key sarcopenia marker.
Change from Baseline in Short Physical Performance Battery (SPPB) Score at 6 Months | Baseline (Month 0) to Month 6
  Composite score from balance tests, 4-meter gait speed, and chair rise test. Score ranges from 0 to 12, with ≤8 indicating poor physical performance.
Change from Baseline in Gait Speed (4-Meter Walk Test) at 6 Months | Baseline (Month 0) to Month 6
  Average walking speed over 4 meters. Lower speeds (<0.8 m/s) are associated with higher frailty and fall risk.
Change from Baseline in Timed Up and Go (TUG) Test Performance at 6 Months | Baseline (Month 0) to Month 6
  Time to rise from a chair, walk 3 meters, turn, return, and sit. Times ≥13.5 seconds indicate increased fall risk.
Change from Baseline in Estimated Skeletal Muscle Mass Index at 6 Months | Baseline (Month 0) to Month 6
  Calculated using anthropometric data via Lee et al.'s validated formula.
Change in Rectus Femoris and Vastus Lateralis Muscle Thickness at 6 Months | Baseline (Month 0) to Month 6
  Ultrasound-based assessment of muscle thickness and adipose tissue content in the dominant lower limb.
Change from Baseline in Mini Nutritional Assessment-Short Form (MNA-SF) Score at 6 Months | Baseline (Month 0) to Month 6
  Nutrition screening tool (score 0-14). Categories: well-nourished (>11), at risk (8-11), malnourished (<8).
Change from Baseline in Mini-Mental State Examination (MMSE) Score at 6 Months | Baseline (Month 0) to Month 6
  Cognitive status measured with MMSE (score 0-30). Scores <26 suggest cognitive impairment.
Number of Participants with Hospital Admissions During the Study Period | Baseline (Month 0) to Month 6
  Self-reported or caregiver-reported data on hospitalizations.
Number of Participants Reporting Falls During the Study Period | Baseline (Month 0) to Month 6
  Number of self-reported falls tracked throughout the study.
Adherence to Home-Based Exercise Sessions (Self-Reported Completion Rate) | Over the 12-week intervention
  Percentage of home-based sessions completed, based on self-records and phone follow-up.
Self-Reported Enjoyment of Physical Activity (Likert Scale) at 6 Months | At Month 6
  Degree of enjoyment assessed on a Likert scale from 1 (not enjoyable) to 5 (very enjoyable).